CLINICAL TRIAL: NCT04027946
Title: A Phase II Study of LMB-100 Followed by Pembrolizumab in the Treatment of Adults With Mesothelin-Expressing Non-Squamous Non-Small Cell Lung Cancer (NSCLC)
Brief Title: LMB-100 Followed by Pembrolizumab in the Treatment of Adults With Mesothelin-Expressing Non-Squamous Non-Small Cell Lung Cancer (NSCLC)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated due to slow accrual.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Azam Ghafoor, Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 190127; 19-C-0127
Record Dates: First submitted 2019-07-19; First posted 2019-07-22 (Actual); Results first posted 2023-07-18 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-03

CONDITIONS: Lung Cancer; Non-Small Cell Lung Cancer; Adenocarcinoma of Lung
Keywords: Immunotherapy; Checkpoint Inhibitor; Monoclonal Antibody; Lung Adenocarcinoma
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung | interventions — LMB-100; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Mesothelin Expressing Non-Small Cell Lung Cancer Participants (Experimental): LMB-100 + Pembrolizumab
  Interventions: Drug: LMB-100; Drug: pembrolizumab; Diagnostic Test: Mesothelin Expression; Diagnostic Test: TrueSight Oncology 500

INTERVENTIONS:
Drug: LMB-100 — Participants will receive LMB-100 on days 1, 3 and 5 of a 21-day cycle for up to 2 cycles.
Drug: pembrolizumab — Participants will receive pembrolizumab on day 1 of each subsequent 21-day cycle.
  Other Names: Keytruda
Diagnostic Test: Mesothelin Expression — Testing for mesothelin expression performed at screening
Diagnostic Test: TrueSight Oncology 500 — Testing for ROS oncogene 1 (ROS1) gene, anaplastic lymphoma kinase (ALK) and epidermal growth factor receptor (EGFR) variations performed at screening.

SUMMARY:
Background:

Over 230,000 new lung cancer cases are diagnosed every year in the United States (U.S.) About 80% of lung cancers are non- small cell lung cancer (NSCLC). Most people have a more advanced stage of the disease that doesn't respond well to standard treatment. Researchers want to see if a combination of drugs may be able to help.

Objective:

To find out if LMB-100 followed by pembrolizumab can help tumors to shrink in people with NSCLC.

Eligibility:

People ages 18 and older with NSCLC that has not responded to standard therapies

Design:

Participants will be screened with:

* Medical history
* Physical exam
* Tumor sample. If one is not available, they will have a biopsy.
* Assessments of ability to perform normal activities
* Lung function tests
* Blood, heart, and urine tests
* Computed tomography (CT) and positron emission tomography (PET). They will lie in a machine that takes pictures of the body.

Participants will take LMB-100 in 21-day cycles for up to 2 cycles. They will take the drug by injection into an arm vein on days 1, 3, and 5 of each cycle. They will stay in the hospital 7-10 days each cycle. Then they will get pembrolizumab by injection into an arm vein every 3 weeks for up to 2 years. They may be able to take pembrolizumab an additional year if their cancer gets worse.

Participants will have repeats of the screening tests throughout the study.

About 30 days and 90 days after they stop treatment, participants will have follow-up visits. Then they will have visits every 6-12 weeks. They will be followed for the rest of their life through phone calls and emails.

DETAILED DESCRIPTION:
Background:

* Mesothelin is expressed in approximately half of all lung adenocarcinomas.
* LMB-100 has demonstrated anti-tumor efficacy against several mesothelin expressing tumor models including non-small cell lung cancer (NSCLC). Programmed death ligand 1 (PD-1) is an Ig superfamily member related to cluster of differentiation (CD28) and cluster of differentiation 152 (CTLA-4) that has been shown to negatively regulate antigen receptor signaling upon engagement of its ligands.
* Pembrolizumab, an immunoglobulin G4 (IgG4) monoclonal antagonist antibody to PD-1, is Food and Drug Administration (FDA) approved in the frontline for advanced non-squamous NSCLC as a single agent with high programmed death-ligand 1 (PD-L1) expression [tumor proportion score (TPS) >=50%] or in combination with platinum-based doublet chemotherapy (PD-L1 unselected). It also approved in the second-line for high PDL1 expressing tumors (TPS >=1%).
* Combination treatment with LMB-100 plus pembrolizumab results in greater anti-tumor efficacy in murine lung cancer model.

Objectives:

-To determine the objective response rate of LMB-100 followed by pembrolizumab in the treatment of subjects with mesothelin-expressing non-squamous non-small cell lung cancer (NSCLC) previously treated with immune checkpoint inhibitors.

Eligibility:

* Histologically confirmed locally advanced or metastatic non-squamous, non-small cell lung cancer lacking an EGFR sensitizing mutation, anaplastic lymphoma kinase (ALK) or ROS oncogene 1 (ROS1) gene rearrangement and not amenable to potentially curative surgical resection or chemoradiation.
* Tumor mesothelin expression of at least 25% of tumor cells as determined by the Laboratory of Pathology at the NCI.
* Subjects must have at least progressed after one prior platinum-based doublet chemotherapy AND standard immune checkpoint inhibitor (ICI) with either frontline single-agent pembrolizumab, or in combination with platinum-based doublet chemotherapy, or second-line single-agent nivolumab, pembrolizumab, or atezolizumab.
* Age >= 18 years.

Design:

* This is an open-label, single center phase II study of LMB-100 followed by pembrolizumab in subjects with mesothelin expressing NSCLC who have progressed on standard therapies
* Subjects will receive LMB-100 at the single agent maximum tolerated dose (MTD) (140mg/kg) on days 1, 3 and 5 of a 21-day cycle for up to 2 cycles and pembrolizumab 200 mg on day 1 of cycle 3 of a 21- day cycle (or cycle 2 if disease progression is observed after 1 cycle) onwards until disease progression (on or after pembrolizumab) or intolerable toxicity for a maximum of 2 years (unless second course initiated).
* The total accrual ceiling for the screening will be set at 100 total patients in order to treat 23 subjects.

ELIGIBILITY:
* INCLUSION CRITERIA:

Participants are eligible to be included in the study only if all of the following criteria apply.

* Male and female participants who are at least 18 years of age on the day of signing the informed consent will be enrolled in the study.
* Subjects must have histologically confirmed diagnosis of non-squamous non-small cell lung cancer not amenable to potentially curative treatments (surgical resection, definitive radiation therapy or a combined modality approach) or targeted agents to actionable epidermal growth factor receptor (EGFR) mutations or Anaplastic lymphoma kinase (ALK) or ROS oncogene 1 (ROS1) gene rearrangement and excluding neuroendocrine tumors. Activating Kirsten rat sarcoma viral oncogene homolog (KRAS) mutations are allowed. The diagnosis must be confirmed by the Laboratory of Pathology, Center for Cancer Research (CCR), National Cancer Institute (NCI). Mutation confirmation may be done by referring institutions or by one of the assays in the Protocol.
* Have provided archival tumor tissue sample or newly obtained fresh core or excisional biopsy of a tumor lesion not previously irradiated. Formalin-fixed, paraffin embedded (FFPE) tissue blocks are preferred to slides. Newly obtained biopsies are preferred to archived tissue.
* Histologically confirmed 25% of tumor cells expressing mesothelin as determined by NCI Laboratory of Pathology. Determination can be made using archival tumor tissue or fresh biopsy.
* Have measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST). Lesions in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
* Subjects must have received prior standard of care treatments for locally advanced or metastatic non-small cell lung cancer (NSCLC).
* Patients must be more than 3 weeks out of systemic treatments, such as chemotherapy.
* All acute toxic effects of any prior radiotherapy, chemotherapy, immunotherapy, or surgical procedure must have resolved to Grade less than or equal to 1, except alopecia (any grade) and Grade 2 peripheral neuropathy.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Evaluation of ECOG is to be performed within 7 days prior to start of study therapy.
* Have adequate organ and marrow function as defined below:
* Patients must have normal organ and marrow function as defined below:

  * hemoglobin greater than or equal to 9g/dL or 5.6 mmol/L
  * absolute neutrophil count greater than or equal to 1,500mcL
  * platelets greater than or equal to 100,000/mcL
  * total bilirubin less than or equal to 2.5 x the upper limit of normal range (UNL) OR direct bilirubin less than or equal to ULN for participants with total bilirubin levels of greater than 1.5 X ULN
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) less than or equal to 2.5 x ULN OR less than or equal to 5 x ULN for subjects with metastatic disease to the liver
  * creatinine greater than or equal to 1.5 x ULN OR creatinine clearance greater than or equal to 50 mL/min for participants with creatinine levels greater than 1.5 X ULN
  * International normalized ratio (INR) or prothrombin time (PT) or activated thromboplastin time (aPTT) greater than or equal to 1.5 X ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants
* Must have left ventricular ejection fraction >50%.
* The effects of LMB-100 on the developing human fetus are unknown. For this reason and because anti-PD-1 antibodies such as pembrolizumab are assumed to be teratogenic:

  * A male participant must agree to use contraception during the treatment period and for at least 180 days after the last dose of study treatment and refrain from donating sperm
  * A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

    * Not a woman of childbearing potential (WOCBP) OR
    * A WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 180 days after the last dose of study treatment.
  * Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
  * Ability of subject to understand and the willingness to sign a written informed consent document.
  * Subjects with non-life-threatening immune-related endocrinopathies or adverse events (AEs) reduced to Grade 1 or 0 after withholding immune checkpoint inhibitors (ICI) or medical intervention are eligible as long as the AE resolved within 12 weeks of last dose and not requiring corticosteroids.

EXCULSION CRITERIA:

* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment. Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e., without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment.
* Subjects who have received prior therapy with LMB-100.

Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks prior to start of study therapy.

* Note: Participants must have recovered from all AEs due to previous therapies to <=Grade 1 or baseline. Participants with <=Grade 2 neuropathy may be eligible.
* Note: If participant received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment.

  * Has received prior radiotherapy within 2 weeks of start of study treatment. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 2-week washout is permitted for palliative radiation (<=2 weeks of radiotherapy) to non-CNS disease.
  * Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist(R)) are live attenuated vaccines and are not allowed.
  * Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to start of study therapy.
  * Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g.., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
  * Has a history of (non-infectious) pneumonitis/interstitial lung disease (ILD) that required steroids or has current pneumonitis/ILD
  * Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
  * Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
  * A WOCBP who has a positive urine pregnancy test within 72 hours prior to start of study therapy. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. Note: In the event that 72 hours have elapsed between the screening pregnancy test and the first dose of study treatment, another pregnancy test (urine or serum) must be performed and must be negative in order for subject to start receiving study medication.
  * Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 180 days after the last dose of trial treatment. Pregnant women are excluded from this study because LMB-100 + pembrolizumab are agents with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with LMB-100 + pembrolizumab, breastfeeding should be discontinued if the mother is treated with LMB-100 + pembrolizumab. These potential risks may also apply to other agents used in this study.
  * Has a known history of Human Immunodeficiency Virus (HIV). HIV positive patients will be excluded due to a theoretical concern that the degree of immune suppression associated with the treatment may result in progression of HIV infection. (Note: No HIV testing is required)
  * Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV ribonucleic acid (RNA [qualitative] is detected) infection. or active hepatitis B virus (HBV) or HCV infection. (Note: No testing for Hepatitis B and Hepatitis C is required.)
  * Has a known additional malignancy that is progressing or has required active treatment within the past 2 years. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g., breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.
  * Has an active infection requiring systemic therapy.
  * Participants with contra-indication and/or history of severe hypersensitivity reactions to any components related to LMB-100 or pembrolizumab (or any other immune checkpoint inhibitor such as Programmed death ligand 1 (PD-1), programmed death-ligand 1 (PD-L1) and cluster of differentiation 152 (CTLA-4).
  * Active or uncontrolled infections.
  * Subjects who experienced severe or life-threatening immune-related AEs with prior immune checkpoint therapy requiring medical intervention (steroid or immunosuppressant drugs) and permanent discontinuation of therapy, will be excluded. These include, but not limited to colitis, autoimmune hepatitis, hypophysitis, hyperthyroidism, nephritis, myocarditis, Guillain-Barré syndrome (GBS), encephalitis.
  * Subjects with a history of pneumonitis that required steroids will be excluded.
  * Recruitment Strategies

Information about the study will be posted on sites such as clinicaltrials.gov and the Center for Cancer Research (CCR) recruitment website. Subjects will also be drawn from patients seen at the thoracic clinic at the National Institutes of Health (NIH) Clinical Center as well as from referrals from outside providers. Social media platforms managed by NIH/National Cancer Institute (NCI) may also be used to publicize the study. There is no plan to advertise this study at this time.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-09-11 (Actual); Primary Completion 2020-06-17 (Actual); Study Completion 2023-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Azam Ghafoor, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. In addition, all large-scale genomic sequencing data will be shared with subscribers to the database of Genotypes and Phenotypes (dbGaP).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely. Genomic data are available once genomic data are uploaded per protocol Genomic Data Sharing Plan (GDS) plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to Biomedical Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI). Genomic data are made available via the database of Genotypes and Phenotypes (dbGaP) through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2019-C-0127.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Mesothelin Expressing Non-Small Cell Lung Cancer Participants: LMB-100 + Pembrolizumab
  LMB-100: Participants will receive LMB-100 140mcg/kg on days 1, 3 and 5 of a 21-day cycle for up to 2 cycles.
  Pembrolizumab: Participants will receive 200 mg pembrolizumab on day 1 of each subsequent 21-day cycle for up to 2 years or until disease progression.
  Mesothelin Expression: Testing for mesothelin expression performed at screening.
  TrueSight Oncology 500: Testing for ROS oncogene 1 (ROS1) gene, anaplastic lymphoma kinase (ALK) and epidermal growth factor receptor (EGFR) variations performed at screening.
Period: Overall Study
Arm/Group | Mesothelin Expressing Non-Small Cell Lung Cancer Participants
Started | 6
Completed | 3
Not Completed | 3
Not completed — Screen failures | 3

BASELINE CHARACTERISTICS:
Population: Although 3 participants were screen failures, data collected for all (6) participants enrolled is shown here.
Arm/Group | Mesothelin Expressing Non-Small Cell Lung Cancer Participants
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.12 (7.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With Partial Response or Complete Response Reported With an 80% Confidence Interval
Description: Participants with a partial response or complete response is reported with an 80% confidence interval. Response was evaluated by the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. Complete response is disappearance of all target lesions. Partial response is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters.
Time Frame: End of treatment, an average of 83 days.
Population: 3/6 participants were analyzed because 3 were screen failures.
Measure: Number (80% Confidence Interval); unit: proportion of participants
Arm/Group | Mesothelin Expressing Non-Small Cell Lung Cancer Participants
Number analyzed (Participants) | 3
proportion of participants | 0 [0 to 0]

2. Primary Outcome: Proportion of Participants With Partial Response or Complete Response Reported With an 95% Confidence Interval
Description: Participants with a partial response or complete response is reported with an 95% confidence interval. Response was evaluated by the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. Complete response is disappearance of all target lesions. Partial response is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters.
Time Frame: End of treatment, an average of 83 days.
Population: 3/6 participants were analyzed because 3 were screen failures.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Mesothelin Expressing Non-Small Cell Lung Cancer Participants
Number analyzed (Participants) | 3
proportion of participants | 0 [0 to 0]

3. Secondary Outcome: Overall Response (OR)
Description: The best overall response is the best response recorded from the start of the treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the treatment started). The participant's best response assignment will depend on the achievement of both measurement and confirmation criteria. Response was evaluated by the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. Complete response (CR) is disappearance of all target lesions. Partial response (PR) is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters. Progressive disease (PD) is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study. Stable disease (SD) is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
Time Frame: From the start of the treatment until disease progression/recurrence (taking as reference for progressive disease), an median of 22.9 months.
Population: 3/6 participants were analyzed because 3 were screen failures.
Measure: Count of Participants; unit: Participants
Arm/Group | Mesothelin Expressing Non-Small Cell Lung Cancer Participants
Number analyzed (Participants) | 3
Participants
  Complete Response | 0
  Partial Response | 0
  Stable Disease | 2
  Progressive Disease | 1

4. Secondary Outcome: Number of Participants With a Response
Description: Response was evaluated by the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. Complete response (CR) is disappearance of all target lesions. Partial response (PR) is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters. Progressive disease (PD) is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study. Stable disease (SD) is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
Time Frame: Beginning at the date a participant is noted to have at least a partial response (PR), an average of 2.7 months.
Population: 3/6 participants were analyzed because 3 were screen failures.
Measure: Count of Participants; unit: Participants
Arm/Group | Mesothelin Expressing Non-Small Cell Lung Cancer Participants
Number analyzed (Participants) | 3
Participants
  Complete Response | 0
  Partial Response | 0
  Stable Disease | 2
  Progressive Disease | 1

5. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression free survival (PFS) is defined as the duration of time from start of treatment to time of progression (on or after pembrolizumab) or death, whichever occurs first, calculated from the on-study date using the Kaplan-Meier method.
Time Frame: Time from start of treatment to time of progression (on or after pembrolizumab) or death, whichever occurs first, calculated from the on-study date using the Kaplan-Meier method, an average of 2.7 months.
Population: 3/6 participants were analyzed because 3 were screen failures.
Measure: Median (Full Range); unit: Months
Arm/Group | Mesothelin Expressing Non-Small Cell Lung Cancer Participants
Number analyzed (Participants) | 3
Months | 3.0 [3 to 4.3]

6. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the duration of time from start of treatment to death from any cause.
Time Frame: Time from the start of treatment to death from any cause, a median of 22.9 months
Measure: Median (Full Range); unit: Months
Arm/Group | Mesothelin Expressing Non-Small Cell Lung Cancer Participants
Number analyzed (Participants) | 3
Months | 22.9 [3.2 to 39.3]

7. Secondary Outcome: Proportion of Participants With Grade 3 and Grade 4 Adverse Events Possibly, Probably, and Definitely Related to LMB-100
Description: Adverse events were evaluated according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Grade 3 is severe. Grade 4 is life-threatening.
Time Frame: Date treatment consent signed to date off study, approximately 48.7 months
Population: 3/6 participants were analyzed because 3 were screen failures.
Measure: Number; unit: proportion of participants
Groups:
- Grade 3 Possibly Related; Grade 3 Probably Related; Grade 3 Definitely Related: Grade 3 is severe.
- Grade 4 Possibly Related; Grade 4 Probably Related; Grade 4 Definitely Related: Grade 4 is life- threatening.
Arm/Group | Grade 3 Possibly Related | Grade 3 Probably Related | Grade 3 Definitely Related | Grade 4 Possibly Related | Grade 4 Probably Related | Grade 4 Definitely Related
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3
proportion of participants | 0 | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Proportion of Participants With Grade 3 and Grade 4 Adverse Events Possibly, Probably, and Definitely Related to Pembrolizumab
Description: as for outcome 7
Time Frame: Date treatment consent signed to date off study, approximately 48.7 months
Measure: Number; unit: proportion of participants
Arm/Group | Grade 3 Possibly Related | Grade 3 Probably Related | Grade 3 Definitely Related | Grade 4 Possibly Related | Grade 4 Probably Related | Grade 4 Definitely Related
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3
proportion of participants | 0 | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Number of Participants Who Are Treated Who Are Unable to Tolerate the Treatment Other Than Development of Adverse Events
Description: Participants who are treated who are unable to tolerate the treatment other than development of adverse events
Time Frame: Date treatment consent signed to date off study, approximately 48.7 months
Population: 3/6 participants were analyzed because 3 were screen failures.
Measure: Count of Participants; unit: Participants
Arm/Group | Mesothelin Expressing Non-Small Cell Lung Cancer Participants
Number analyzed (Participants) | 3
Participants | 0

10. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0)
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 48.7 months
Measure: Count of Participants; unit: Participants
Arm/Group | Mesothelin Expressing Non-Small Cell Lung Cancer Participants
Number analyzed (Participants) | 3
Participants | 3

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 48.7 months.
Description: 3/6 participants were analyzed because 3 were screen failures. There were 3 deaths due to progression and not related to the study.
Arm/Group | Mesothelin Expressing Non-Small Cell Lung Cancer Participants
All-Cause Mortality (participants affected / at risk) | 3/3
Serious Adverse Events (participants affected / at risk) | 3/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mesothelin Expressing Non-Small Cell Lung Cancer Participants (N=3)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Hepatocellular carcinoma - secondary malignancy
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mesothelin Expressing Non-Small Cell Lung Cancer Participants (N=3)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 2 (2)
Alanine aminotransferase increased (Investigations) | 1 (2)
Anemia (Blood and lymphatic system disorders) | 3 (11)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 2 (3)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 1 (1)
CPK increased (Investigations) | 1 (1)
Capillary leak syndrome (Vascular disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (6)
Edema limbs (General disorders) | 1 (1)
Electrocardiogram QT corrected interval prolonged (Cardiac disorders) | 1 (1)
Eye pain (Eye disorders) | 1 (1)
Fatigue (General disorders) | 2 (4)
Fever (General disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Hematuria (Renal and urinary disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (9)
Hypokalemia (Metabolism and nutrition disorders) | 1 (4)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 3 (5)
Hypotension (Vascular disorders) | 2 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Lymphocyte count decreased (Investigations) | 3 (7)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Pain (General disorders) | 1 (5)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Proteinuria (Renal and urinary disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 3 (7)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Thrush (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Weight gain (Investigations) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (4):
  • Study Protocol and Statistical Analysis Plan (2021-12-03): https://cdn.clinicaltrials.gov/large-docs/46/NCT04027946/Prot_SAP_000.pdf
  • Informed Consent Form: Screening Consent (2020-01-28): https://cdn.clinicaltrials.gov/large-docs/46/NCT04027946/ICF_001.pdf
  • Informed Consent Form: Affected Patients Consent (2021-12-21): https://cdn.clinicaltrials.gov/large-docs/46/NCT04027946/ICF_002.pdf
  • Informed Consent Form: Treatment After Progression Consent (2020-01-28): https://cdn.clinicaltrials.gov/large-docs/46/NCT04027946/ICF_003.pdf